CLINICAL TRIAL: NCT01741259
Title: A Comparison of Meperidine for Post-Cesarean Analgesia: Bolus Versus Infusion and Bolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Christy L Morgan, MD, Obstetric Anesthesiologist, Mercy Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 371047-1
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Cesarean Section
Keywords: analgesia; meperidine; epidural
MeSH Terms: conditions — Agnosia | interventions — Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meperidine PCEA (Experimental): Epidural Meperidine (5mg/ml) bolus of 20 mg, lockout of 30 min, hourly limit of 50 mg.
  Interventions: Drug: Meperidine
- Meperidine PCEA with basal (Experimental): Epidural meperidine (5mg/ml) basal rate of 10 mg/hr, bolus 20 mg, lockout 30 min, hourly limit 40 mg
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: Meperidine
  Other Names: Demerol

SUMMARY:
The purpose of this study is to determine if epidural meperidine administered by patient-controlled bolus button is equivalent to a low dose infusion plus patient-controlled bolus.

DETAILED DESCRIPTION:
The objective of this study is to compare the efficacy, patient satisfaction, and incidence of side effects of meperidine patient-controlled epidural analgesia (PCEA) with and without a basal infusion for post-cesarean section analgesia.

ELIGIBILITY:
Inclusion Criteria are as follows:

* Over the age of 18
* Undergoing non-urgent, non-emergent cesarean section at Mercy Hospital St. Louis

Exclusion Criteria:

* non-English speaking
* mentally disabled
* allergy to meperidine
* seizure disorder
* renal impairment defined as a serum creatinine >0.8 mg/dL or patients who give a history of renal impairment
* fever greater than 101
* patients receiving low molecular weight heparin at any dose or unfractionated heparin at doses greater than 5000 u subcutaneous twice daily
* pre-eclampsia requiring magnesium due to post-partum room assignment
* obstructive sleep apnea due to post-partum room assignment
* post-partum hemorrhage due to post-partum room assignment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy L Morgan, MD, Principal Investigator — Mercy Hospital St. Louis
Locations (1):
- Mercy Hospital St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 Patients were excluded after enrollment but prior to randomization. 3 were due to not having an epidural in place after surgery - 2 had accidental intrathecal catheter placement and 1 was to be started on lovenox. Another had a missing consent form and the other was started on magnesium sulfate which was an exclusion criterion.
Groups:
- Meperidine PCEA: Epidural Meperidine (5mg/ml) bolus of 20 mg, lockout of 30 min, hourly limit of 50 mg.
  Meperidine
- Meperidine PCEA With Basal: Epidural meperidine (5mg/ml) basal rate of 10 mg/hr, bolus 20 mg, lockout 30 min, hourly limit 40 mg
  Meperidine
Period: Overall Study
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Started | 133 | 135
Completed | 127 | 129
Not Completed | 6 | 6
Not completed — Protocol Violation | 6 | 4
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal | Total
Number analyzed (Participants) | 127 | 129 | 256
Age, Continuous [Median (Standard Deviation); unit: years] | 31 (4.39) | 31 (4.81) | 31 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 129 | 256
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 129 | 256
Primary vs repeat Cesarean Section [Count of Participants; unit: Participants]
  Primary CS | 37 | 41 | 78
  Repeat CS | 90 | 88 | 178
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.03 (7.22) | 32.18 (6.17) | 33.09 (6.76)

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Score With Movement
Description: Verbal Pain Score on a 0-10 scale is recorded by the nurse at 0, 4, 8, 12, 16, 20, 24, 28, 32, 36,40, 44, and 48 hours after transfer to the post-partum floor. On this scale, 0 represents no pain at all and 10 represents the worst pain imaginable. Because we were relying on nurses to capture this data in the course of normal patient care, scores within 1 hour before or after the goal time were accepted. For each patient, the average of all pain scores was taken and this was considered to be the average pain score while the epidural meperidine was being given.
Time Frame: 36-48 hours post-op (until epidural is stopped)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
units on a scale | 1.92 (1.00) | 1.50 (1.06)

2. Secondary Outcome: Nausea and Vomiting
Description: The incidence of nausea and vomiting will be estimated by the administration of ondansetron during the study period as recorded in the patient record.
Time Frame: 36-48 hours post-op (until epidural is stopped)
Measure: Number; unit: participants
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
participants | 1 | 3

3. Secondary Outcome: Pruritus
Description: The incidence of pruritus will be estimated by the administration of diphenhydramine or nalbuphine during the study period as recorded in the patient record.
Time Frame: 36-48 hours post-op (until the epidural is stopped)
Measure: Number; unit: participants
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
participants | 20 | 10

4. Secondary Outcome: Dysphoria
Description: The incidence of dysphoria will be captured when a nurse calls the anesthesia team to alert them. This information is tracked on the physician rounding sheet. The record will also be reviewed if an epidural is discontinued earlier than the morning of the second post-operative day to find out if dysphoria was the cause.
Time Frame: 36-48 hours post-op (until epidural is stopped)
Measure: Number; unit: participants
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
participants | 0 | 0

5. Secondary Outcome: Inadequate Analgesia
Description: Patients routinely get scheduled ibuprofen as an adjunct to the epidural infusion. The record will be reviewed to see if ketorolac is substituted for ibuprofen or other pain medications such as acetaminophen either alone or in combination with oxycodone or other narcotic pain relievers are administered. The record will also be reviewed if an epidural is discontinued earlier than the morning of the second post-operative day to find out if inadequate analgesia was the cause.
Time Frame: 36-48 hours post-op (until the epidural is stopped)
Measure: Number; unit: participants
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
participants | 7 | 3

6. Secondary Outcome: Adverse Outcomes
Description: Adverse outcomes such as seizures or respiratory depression will be reported to anesthesia personnel by nursing if they occur. Patients are monitored for respiratory rate and sedation every 1 hour for 24 hours, then every 2 hours for 24 hours. Pulse, blood pressure, and neurocirculatory checks are performed every 2 hours for 24 hours and then every 4 hours per our nursing protocol.
Time Frame: 36-48 hours post-op (until the epidural is stopped)
Measure: Number; unit: participants
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
participants | 0 | 0

7. Secondary Outcome: Total Drug Dose
Description: Pharmacy will generate a report of the drug total from the pump on return to pharmacy.
Time Frame: 48 hours post-op or when the epidural is stopped
Measure: Mean (Standard Deviation); unit: milligrams of drug per hour
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 127 | 129
milligrams of drug per hour | 5.42 (2.28) | 8.49 (4.19)

8. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #1
Description: Please indicate on 0-10 scale the least pain you had in first 24 hours. 0 represents no pain and 10 represents the worst pain possible. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 1.89 (.152) | 1.45 (.153)

9. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #2
Description: On 0-10 scale, indicate the worst pain you had in first 24 hours. 0 represents no pain and 10 represents the worst pain possible. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 5.79 (.175) | 5.10 (.199)

10. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #3
Description: How often were you in severe pain in the first 24 hours (percentage 0-100%). 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
percentage of time | 14.47 (1.778) | 11.78 (1.327)

11. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #4a
Description: How much, on 0-10 scale, did pain interfere with doing activities in bed (turning, sitting up, repositioning) where 0 is does not interfere and 10 is completely interferes. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 121 | 117
units on a scale | 4.04 (.222) | 3.13 (.203)

12. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #4b
Description: How much, on a 0-10 scale, did pain interfere with doing activities out of bed (walking, sitting in chair, standing at sink) where 0 is does not interfere and 10 is completely interferes. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 120 | 114
units on a scale | 4.02 (.235) | 3.71 (.238)

13. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #4c
Description: How much, on a 0-10 scale, did pain interfere with falling asleep where 0 is does not interfere and 10 is completely interferes. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 2.016 (.2171) | 1.487 (.1853)

14. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #4d
Description: How much, on a scale of 0-10, did pain interfere with staying asleep where 0 is does not interfere and 10 is completely interferes. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 117
units on a scale | 2.04 (.210) | 1.68 (.210)

15. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #5a
Description: On a scale of 0-10, how much did the pain cause you to feel anxious where 0 is not at all anxious and 10 is extremely anxious. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 1.311 (.1965) | 1.504 (.1808)

16. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #5b
Description: On a scale of 0-10, how much did pain cause you to feel depressed where 0 is not al all and 10 is extremely. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 117
units on a scale | .47 (.123) | .34 (.092)

17. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #5c
Description: How much, on a scale of 0-10, did the pain cause you to feel frightened where 0 is not at all and 10 is extremely. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 117
units on a scale | .85 (.171) | .79 (.154)

18. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #5d
Description: How much, on a scale of 0-10, did the pain cause you to feel helpless where 0 is not at all and 10 is extremely. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 117
units on a scale | 1.42 (.227) | 1.49 (.220)

19. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #6a
Description: On a scale of 0-10, what was the severity of your nausea where 0 is none and 10 is severe. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | .49 (.110) | .69 (.143)

20. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #6b
Description: On a 0-10 scale, how severe was your drowsiness where 0 is none and 10 is severe. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 2.26 (.211) | 2.91 (.231)

21. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #6c
Description: On a 0-10 scale, how severe was your itching where 0 is none and 10 is severe. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 121 | 118
units on a scale | 2.661 (.2557) | 2.419 (.2537)

22. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #6d
Description: On a 0-10 scale, how severe was your dizziness where 0 is not at all and 10 is extremely. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | .84 (.152) | 1.13 (.176)

23. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #7
Description: Select the percentage (from 0%-100%) of pain relief you received from all medical and non-medical treatments in the first 24 hours. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: percentage of pain relieved
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
percentage of pain relieved | 77.05 (1.733) | 81.82 (1.592)

24. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #8
Description: On a 0-10 scale, were you allowed to participate in decisions about your pain treatment as much as you wanted to with 0 being not at all and 10 being entirely. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 8.996 (.1932) | 9.258 (.1547)

25. Secondary Outcome: American Pain Society Patient Outcome Questionnaire #9
Description: On a 0-10 scale, how satisfied are you with the results of your pain treatment with 0 being extremely dissatisfied and 10 being extremely satisfied. 122 patients in the Meperidine PCEA no basal group completed their questionnaires while 118 in the Meperidine PCEA with basal group completed a questionnaire. Some patients did not answer all the questions on the questionnaire, if a question was left blank, it was not analyzed for that patient but the rest of the questionnaire was included.
Time Frame: Survey day epidural stopped
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
Number analyzed (Participants) | 122 | 118
units on a scale | 8.76 (.183) | 9.41 (.106)

ADVERSE EVENTS:
Time Frame: Until discharge from hospital (usually 4 days post cesarean section)
Arm/Group | Meperidine PCEA | Meperidine PCEA With Basal
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/129
Other Adverse Events (participants affected / at risk) | 0/127 | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No